CLINICAL TRIAL: NCT01157845
Title: Use of the BreathID Methacetin Breath Test to Assess Hepatic Metabolic Reserve and to Predict Hepatic Decompensation in Patients Awaiting Liver Transplantation
Brief Title: Use of Methacetin Breath Test to Predict Liver Failure in Patients With Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Meridian Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VirginiaCU HM12041
Record Dates: First submitted 2010-07-02; First posted 2010-07-07 (Estimated); Results first posted 2014-03-04 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-04

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laboratory assay (Experimental)
  Interventions: Device: BreathID (Methacetin breath test)

INTERVENTIONS:
Device: BreathID (Methacetin breath test) — 13C-labeled methacetin (75 mg) is given to the patient by mouth in a small volume of water, and expired 13C-labeled carbon dioxide is measured from a nasal cannula.
  Other Names: BreathID (Exalenz Bioscience LTD)

SUMMARY:
The methacetin breath test (MBT) is a non-invasive liver function test which measures the ability of the liver to metabolize a tracer dose of a compound to carbon dioxide, which is exhaled. The study hypothesis is that measurement of the MBT will allow earlier detection of a decline in liver function in patients with cirrhosis who are awaiting liver transplantation.

ELIGIBILITY:
Inclusion criteria:

1. Being considered for placement or already on the liver transplantation waiting list
2. Cirrhosis caused by any cause of chronic liver disease.
3. Age > 18 years

Exclusion criteria:

1. Known or suspected hepatocellular carcinoma
2. Prior TIPS placement
3. Severe congestive heart failure
4. Severe pulmonary hypertension
5. Uncontrolled diabetes mellitus (HBA1C >9.5%)
6. Any autoimmune disorder, which is currently being treated with prednisone or any other immune suppressive medication.
7. Previous surgical bypass surgery for morbid obesity (BMI >45)
8. Extensive small bowel resection
9. Patients currently receiving total parenteral nutrition if they have contraindications to oral drugs
10. Women who are pregnant
11. Patients who are allergic to acetaminophen/ paracetamol or any other related medications
12. Patients with an acute current exacerbation of chronic obstructive pulmonary disease or bronchial asthma.
13. Patients that are taking hepatotoxin drugs
14. Patient, based on the opinion of the investigator, should not be enrolled into this study
15. Patient is unable or unwilling to sign informed consent.
16. Patients that are participating in other clinical trials evaluating experimental treatments or procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2010-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Stravitz, MD, Principal Investigator — Virginia Commonwealth University
Locations (4):
- United States (3):
  - Henry Ford Health System, Detroit, Michigan
  - Medical University of South Carolina, Charleston, South Carolina
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
- Hadassah Medical Center, Jerusalem, Israel, Israel

REFERENCES:
- [Background] Braden B, Faust D, Sarrazin U, Zeuzem S, Dietrich CF, Caspary WF, Sarrazin C. 13C-methacetin breath test as liver function test in patients with chronic hepatitis C virus infection. Aliment Pharmacol Ther. 2005 Jan 15;21(2):179-85. doi: 10.1111/j.1365-2036.2005.02317.x. PMID 15679768

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Laboratory Assay
Started | 165
Completed | 130
Not Completed | 35
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 12
Not completed — Physician Decision | 3
Not completed — Protocol Violation | 13
Not completed — Study was ended | 1
Not completed — Device malfunction | 1

BASELINE CHARACTERISTICS:
Population: All chronic liver disease patients with clinically proven cirrhosis and candidates for liver transplant.
Arm/Group | Laboratory Assay
Number analyzed (Participants) | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (10.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 163
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 99
  Israel | 66
Chronic Liver Disease Etiology [Number; unit: participants]
  Alcoholic Liver Disease | 22
  Cholestatic | 16
  Cryptogenic cirrhosis | 17
  Hepatitis B | 5
  Hepatitis C | 75
  Fatty LIver | 19
  Other | 11

OUTCOME MEASURES:

1. Primary Outcome: Mortality From Liver Failure
Description: Patient dies of liver-related causes within 1 year of study entry
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Laboratory Assay
Number analyzed (Participants) | 165
participants | 11

2. Secondary Outcome: Liver Transplantation
Description: Patient experiences complications of liver failure within 1 year of study entry and undergoes liver transplantation
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Laboratory Assay
Number analyzed (Participants) | 165
participants | 34

ADVERSE EVENTS:
Description: No breath test related adverse events reported.
Arm/Group | Laboratory Assay
Serious Adverse Events (participants affected / at risk) | 107/165
Other Adverse Events (participants affected / at risk) | 92/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laboratory Assay (N=165)
Transplantation (Hepatobiliary disorders) | 34 (34) — Patients in this trial are candidates for liver transplant. When there is a sudden change for the worse in their condition, they may be prioritized for transplantation/
Death (Hepatobiliary disorders) | 11 (11) — Some patients waiting for a liver transplant will die before they find a matching liver
Abdominal pain (Hepatobiliary disorders) | 8 (11) — Indirectly related- to- liver ailments may occur in patients with advanced liver disease.
Hepatic Encephelopathy (Hepatobiliary disorders) | 6 (13) — Lack in full cognitive abilities is common in patients with advanced liver disease.
Ascites (Hepatobiliary disorders) | 5 (6) — Ascites ( collection of fluid) is common in patients with advanced liver disease
GI Bleeding (Hepatobiliary disorders) | 5 (5) — GI bleeding (varices) is common in patients with advanced liver disease
Liver related procedure-TIPS (Surgical and medical procedures) | 5 (5) — The patients with advanced liver disease are occasionally hospitalized for preventative treatments such as TIPS (Transjugular intrahepatic portosystemic shunt)
SBP (spontaneous bacterial peritonitis) (Hepatobiliary disorders) | 8 (13) — Common in advanced cirrhotics
Renal failure (Renal and urinary disorders) | 5 (6) — The lack of liver functionality in cirrhotic patients may lead to certain severe events such as renal failure
Cellulitis (Hepatobiliary disorders) | 2 (2)
Fluid in respiratory tract (Hepatobiliary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Hyponatremia (Blood and lymphatic system disorders) | 3 (3)
Bowel Resection (Gastrointestinal disorders) | 1 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Band Ligation Procedure (Surgical and medical procedures) | 2 (2) — The patients with advanced liver disease are occasionally hospitalized for preventative treatments such as band ligation
RFA (Surgical and medical procedures) | 1 (1) — The patients with advanced liver disease are occasionally hospitalized for preventative treatments such as RFA (radio frequency ablation)
Sepsis (Infections and infestations) | 7 (9) — The lack of liver functionality in cirrhotic patients may lead to certain severe events such as sepsis
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laboratory Assay (N=165)
Diarrhea (Gastrointestinal disorders) | 8 (9)
Hernia (General disorders) | 2 (3)
Abdominal Pain (Gastrointestinal disorders) | 5 (16)
Assorted Pains (excluding abdominal) (General disorders) | 13 (19)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hip Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Headaches, Migraines, Dizziness (Nervous system disorders) | 6 (12)
Fatigue (General disorders) | 3 (3)
Blood related disorders (Blood and lymphatic system disorders) | 5 (5)
Infections (Infections and infestations) | 5 (5) — Various infections not liver related and not specified
Depression (Psychiatric disorders) | 3 (3)
Out-patient procedure-Paracentesis (Surgical and medical procedures) | 11 (64)
Fluid accumulation-edema (General disorders) | 2 (2)
Malignancies (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Itching (General disorders) | 5 (5)
Others (General disorders) | 6 (6)
Seizure (Nervous system disorders) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hip replacement (Musculoskeletal and connective tissue disorders) | 1 (1)
Difficulty ambulating (Musculoskeletal and connective tissue disorders) | 2 (2)
Melena (Gastrointestinal disorders) | 1 (1)
Other Gastrointestinal Disorders (Gastrointestinal disorders) | 1 (1) — Non-specified disorders
Lightheadedness (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Suicidal thoughts (Psychiatric disorders) | 1 (1)
Other psychiatric disorders (Psychiatric disorders) | 1 (1) — Unspecified psychiatric disorders
Pleural Effusion (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less